CLINICAL TRIAL: NCT01328015
Title: The Use of Oxybutynin in Women After Thoracoscopic Sympathectomy and the Effect on Plantar Hyperhidrosis
Brief Title: A Study to Compare Oxybutynin to a Placebo in Women and the Effect on Plantar Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Altair da Silva Costa Junior, Federal University of São Paulo - Thoracic surgery departament
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Oxybutynin and Hyperhidrosis
Record Dates: First submitted 2011-03-29; First posted 2011-04-04 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2010-11

CONDITIONS: Hyperhidrosis
Keywords: hyperhidrosis; oxybutynin; plantar sweating; compensatory sweating
MeSH Terms: conditions — Hyperhidrosis | interventions — oxybutynin; Cholinergic Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxybuynin, hyperhidrosis (Active Comparator)
  Interventions: Drug: Oxybutynin 5 mg pills
- placebo - sugar pill (Placebo Comparator)
  Interventions: Drug: Oxybutynin 5 mg pills

INTERVENTIONS:
Drug: Oxybutynin 5 mg pills — ½ pill oral 12/12h for 3 days
  01 ½ pills oral morning and evening for 3 days Continue 1 pill oral 2x/day for three weeks.
  Other Names: anticholinergic drugs

SUMMARY:
A study in which the experimental treatment procedure is compared to a standard (control) treatment, The use of oxybutynin in the late postoperative thoracic sympathectomy for women:

1. To Evaluate the effect of oxybutynin on plantar hyperhidrosis.
2. To evaluate the effect of oxybutynin in compensatory hyperhidrosis.
3. To compare the results of questionnaires on quality of life and specific for hyperhidrosis to the results of TEWL.

DETAILED DESCRIPTION:
Sweating is the most important mechanism of the body to regulate body temperature, kept at around 36ºC. The thermoregulatory center in the hypothalamus captures data from the blood that passes through the brain and also the receptors of the skin. Sweat is a response to thermal variation, but may also appear in situations of anxiety and stress. The sweating occurs at rest in ambient temperatures greater than 24ºC.

The sweat glands are in greater numbers are located on the palms, soles, face and underarms. Specifically, these regions, such glands are also influenced by psychological factors, different glands located on the back and abdomen that respond to heat.

The hyperhidrosis is a relatively common disorder, affecting between 0.6 to 1% of the population. It is characterized by increased sweat in certain areas of the body such as hands, face, feet and armpits. More frequent in young adults and adolescents, mostly females. This is not a serious illness as life threatening, but this situation is very uncomfortable, causing deep embarrassment social relationships and psychological disorders in the carrier, which often isolate themselves socially and acquire habits that conceal their problem. Primary hyperhydrosis is the most common indication for the performance of thoracic sympathectomy.

Videothoracoscopic sympathectomy is performed for the treatment of palmar hyperhidrosis, axillary or cranial-facial, with improvement ranging from 80 to 95%. Patients with plantar sweating associated with hyperhidrosis may remain even after the operation. Moreover, the compensatory effect occurs in most patients (70%), with sweat in the abdomen and back, among others.

The plant can alleviate hyperhidrosis after thoracic sympathectomy in 50% of patients, by mechanisms not yet understood. The persistence of this sweat is located a source of frequent complaint postoperatively, spatially specific occasions such as wearing sandals, slippers or going barefoot.

The diagnosis of hyperhidrosis is exclusively clinical, based on complaints of patients and their limitations in different areas - social, labor, emotional and psychological. No need for further examination to determine the existence of the disease. Faced with this, the assessment after any treatment, is also made subjectively, ie based on patient's opinion and especially its degree of satisfaction. In an attempt to improve this kind of response to treatment, specific questionnaires were developed on the most important complaints and more frequent, and these questions before and after treatment. Currently the investigators have several questionnaires to assess the treatment of hyperhidrosis, not the diagnosis.

With technological advances, there were devices used to determine the flow of evaporation of skin - called by capacitance hygrometry analysis of transdermal water loss, known by its acronym in English TEWL. This is currently the most promising method for objective measurement of sweat, also used by cosmetics companies for new product research (31,32). The value is determined in grams per square meter per hour (g/m2/h). Still no data in the literature to define the limits of TEWL and its application in real hyperhidrosis. But studies comparing the questionnaires mainly specific quality of life and objective measures of the amount of sweat and post-treatment

There is no drug class specific use for the treatment of hyperhidrosis. Groups of anticholinergic medications, beta-blockers and psychotropic drugs may lead to a decreased sweating, not satisfactorily and without support in the literature.

Oxybutynin is a parasympatholytics with relaxant effect on bladder detrusor muscle by action on muscarinic antagonist. The classic indication is urinary incontinence.

The use of anticholinergic oral drugs in hyperhidrosis is unknown and the experience with oxybutynin is restricted. The literature supports this assertion, only case reports. Its use is limited in the U.S. and Europe for treatment of hyperhidrosis. Even without consensus, it is common to the administration of oxybutynin for the treatment of hyperhidrosis, in empirical and based on personal knowledge.

Objective:

To evaluate the efficacy of oxybutynin in the treatment of plantar hyperhidrosis and its impact on quality of life in women already done thoracic sympathectomy.

Method The sample population will be selected by telephone and/or e-mail from patients in late postoperative (more than six months) of thoracic sympathectomy.

Method of evaluation and research:

Specific questionnaire for plantar hyperhidrosis Questionnaire of quality of life for hyperhidrosis Measurement of sweating with TEWL.

Evaluations will be held before the division of the groups and after four weeks of treatment. The data will be collected: age, length of postoperative BMI and side effects to the medication.

Patients will be divided into two groups - placebo and oxybutynin group. Study randomized clinical trial with placebo. The intervention will be the use of oxybutynin for four weeks at dosage below:

Dosage:

½ cp oral 12/12h for 3 days

01 ½ cp oral morning and evening for 3 days Continue 1 cp oral 2x/day for three weeks. Besides the focus on planting hyperhidrosis, compensatory sweating also evaluate with the same parameters, this being the secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* women with persistent plantar hyperhidrosis with limitation to their usual activities.

Exclusion Criteria:

* pregnancy,
* breastfeeding,
* glaucoma,
* use of tricyclic medications,
* prior use of anticholinergic
* side effects exacerbated, such as diarrhea, gastritis, constipation or dry mouth.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of oxybutynin in plantar hyperhidrosis | 60 days
  Apply the questionnaires of quality of life, specific ones for hyperhidrosis and TEWL before in patients with persistence of plantar sweating after thoracic sympathectomy. After continuous use of oxybutynin for a month, repeated them for comparison.

SECONDARY OUTCOMES:
To evaluate the effect of oxybutynin in compensatory hyperhidrosis | 60 days
  Apply the questionnaires of quality of life, specific ones for hyperhidrosis and TEWL before in patients with persistence of plantar sweating after thoracic sympathectomy. After continuous use of oxybutynin for a month, repeated them for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Altair S Costa Jr, MD, Principal Investigator — Federal University of São Paulo

REFERENCES:
- [Background] Tupker RA, Harmsze AM, Deneer VH. Oxybutynin therapy for generalized hyperhidrosis. Arch Dermatol. 2006 Aug;142(8):1065-6. doi: 10.1001/archderm.142.8.1065. No abstract available. PMID 16924061
- [Background] Mijnhout GS, Kloosterman H, Simsek S, Strack van Schijndel RJ, Netelenbos JC. Oxybutynin: dry days for patients with hyperhidrosis. Neth J Med. 2006 Oct;64(9):326-8. PMID 17057269
- [Derived] Costa Ada S Jr, Leao LE, Succi JE, Perfeito JA, Filho Castelo A, Rymkiewicz E, Filho Aurelio Marchetti M. Randomized trial - oxybutynin for treatment of persistent plantar hyperhidrosis in women after sympathectomy. Clinics (Sao Paulo). 2014 Feb;69(2):101-5. doi: 10.6061/clinics/2014(02)05. PMID 24519200